CLINICAL TRIAL: NCT03500003
Title: Metabolic Signatures Resulting From Acute (Postprandial) Ingestion of Yoghurt or Milk in Humans: Effect of Age
Brief Title: Metabolic Signatures of Dairy Products Ingestion in Humans: Effect of Age
Acronym: FermentoMilk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sergio Polakof (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Agroscope Liebefeld-Posieux Research Station ALP (Other)
Responsible Party: Sponsor-Investigator, Sergio Polakof, PhD, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Organization: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FermentoMilk
Record Dates: First submitted 2018-03-27; First posted 2018-04-17 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Nutrition
Keywords: dairy products; milk; yogurt; metabolomics; elderly

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milk acute intake (Experimental): 14 adult and 14 elderly volunteers will consume 600mL of milk. Blood (11 sampling points) and urine samples (3 collection points) will be collected before the ingestion and during the postprandial period (6h).
  Interventions: Other: Acute milk intake
- Yogurt acute intake (Experimental): 14 adult and 14 elderly volunteers will consume 600mL of yogurt. Blood (11 sampling points) and urine samples (3 collection points) will be collected before the ingestion and during the postprandial period (6h).
  Interventions: Other: Acute Yogurt intake

INTERVENTIONS:
Other: Acute milk intake — Food matrix: milk
  Arms: Milk acute intake
Other: Acute Yogurt intake — Food matrix: yogurt
  Arms: Yogurt acute intake

SUMMARY:
Despite the fact that dairy products are greatly consumed, it remains today very difficult to determine with a classical blood biochemical test whether a person has ingested a fresh fermented dairy product or just milk, while their biological, metabolic and health impacts may be different.

The metabolic footprint left by the consumption of these products could be modified by the age of the consumer. Indeed, in the elderly, the processes of digestion, assimilation and metabolism are known to be altered /different compared to healthy adults. Thus, different metabolic signatures in the elderly could appear as the result of a less effective use and metabolism of the nutrients ingested. This could further also result in different or altered biological effects on dairy products.

DETAILED DESCRIPTION:
The two main objectives of this project are to:

* Determine precisely the plasma and urine metabolic signatures resulting from acute (postprandial) ingestion of yogurt or milk.
* Characterize the metabolic signature following the consumption of these dairy products in the elderly and compared with the signature of reference (adult).
* Understand the mechanisms and metabolic pathways involved if discriminating metabolites between age are detected..

The clinical study is open, monocentric, controlled and randomized, in a cross experimental design.

The study is not performed in a double blind way. However, the measure bias will be limited because of the standardized and objective characteristic of the main criteria. Moreover, biological samples will be analyzed by the same partners of the project. Each subject will be its own control, so that confusion factors related to individual variability will be eliminated.

A total of 28 volunteers (men) will participate in the study: 14 adults and 14 old people (>65 yrs-old). After 3 weeks of controlled diet (without consumption of dairy products) the volunteers will ingest 600g of milk or yogurt. After 1 week of wash-out, the other product will be consumed. Blood and urine will be collected during the postprandial period.

The monocentric characteristic of the study, the low number of subjects and the expertise of the involved staff will enable to limit the number of missing data.

The randomization (latin square) has been established by a bio-statistician of the project before the study started. A document describing the randomization proceeding is confidentially kept.

ELIGIBILITY:
Inclusion Criteria:

* no pathology and no medical treatment
* BMI >=21 and <=30 kg/m²
* normal biological status
* no dislike for diary intake

Exclusion Criteria:

* smoking
* no pathology and no medical treatment (no antibiotics in the last 3 months)
* consumption of nutritional supplements several times at week

Ages: 25 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
Metabolomics: discovery of novel biomarkers of acute dairy intake (milk and yogurt) | Baseline, then ten times during the 6h following product intake on two different days (one milk, one yogurt)
  Analysis of the urine and plasma metabolome

SECONDARY OUTCOMES:
glucose homeostasis markers | Baseline, then ten times during the 6h following product intake on two different days (one milk, one yogurt)
  Analysis of blood glucose and insulin levels
lipid homeostasis markers | Baseline, then ten times during the 6h following product intake on two different days (one milk, one yogurt)
  Analysis of blood cholesterol and triglycerides levels
Inflammation markers | Baseline, then ten times during the 6h following product intake on two different days (one milk, one yogurt)
  IL-6, TNF-alpha blood levels

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine d'Auvergne, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided
The identified individual participant data for all outcome measures will be made available, only after joined consent of promotor and investigator. Data use and transfer to a third party will be performed according to the agreement signed as part of the grant funded by CNIEL.